CLINICAL TRIAL: NCT07189923
Title: Efficacy and Safety of Ablative Fractional CO2 Laser and Platelet-rich Plasma (PRP) With Microneedling for Treatment of Acne Scars: a Real-world Comparative Study
Brief Title: Comparative Real-world Study on Ablative Fractional CO₂ Laser vs PRP With Microneedling for Acne Scar Treatment.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sirajul Islam Medical College (Other)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Azmiree Binte Aslam, Assistant Professor, Department of Dermatology and Venereology, Dr. Sirajul Islam Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/48
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Acne Scars; Ablative Fractional CO₂ Laser Therapy; Platelet-rich Plasma (PRP)
Keywords: Acne Scars; Ablative fractional CO₂ laser therapy; Platelet-rich plasma (PRP); Microneedling; Efficacy; Safety; Bangladesh; Goodman and Baron scale

STUDY DESIGN:
Intervention Model Description: This is a randomized, split-face, open-label trial. Each participant will receive ablative fractional CO₂ laser therapy on one side of the face and platelet-rich plasma (PRP) with microneedling on the other side. The split-face design allows within-participant comparison of the two treatment modalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablative fractional CO2 laser (Active Comparator): Participants will receive ablative fractional CO₂ laser therapy on one side of the face using the SmartXide DOT Fractionated CO₂ Laser system. Treatment parameters include 15 W power, 800 µm spacing, 600 µs dwell time, and stack level 2. A total of three sessions will be administered, each one month apart.
  Interventions: Procedure: Ablative Fractional CO₂ Laser
- Platelet-Rich Plasma (PRP) With Microneedling (Experimental): Participants will receive intradermal injections of autologous PRP followed by microneedling on the opposite side of the face. PRP will be prepared using a double-spin centrifugation method from 8 mL of venous blood. Microneedling will be performed with a Dermapen (12-needle cartridge, 1.5 mm depth) until pinpoint bleeding is observed. A total of three sessions will be administered, each one month apart.
  Interventions: Procedure: Platelet-Rich Plasma (PRP) With Microneedling

INTERVENTIONS:
Procedure: Ablative Fractional CO₂ Laser — Participants will receive ablative fractional CO₂ laser therapy on one side of the face using the SmartXide DOT Fractionated CO₂ Laser system. Treatment parameters: 15 W power, 800 µm spacing, 600 µs dwell time, stack level 2. Sessions: 3, each one month apart.
  Arms: Ablative fractional CO2 laser
Procedure: Platelet-Rich Plasma (PRP) With Microneedling — Participants will receive intradermal autologous PRP injections prepared by double-spin centrifugation from 8 mL of venous blood, followed by microneedling with a Dermapen (12-needle cartridge, 1.5 mm depth). Endpoint: pinpoint bleeding. Sessions: 3, each one month apart.
  Arms: Platelet-Rich Plasma (PRP) With Microneedling

SUMMARY:
Road traffic accidents (RTAs) remain a major public health concern worldwide and in Bangladesh, contributing significantly to injury, disability, and premature death. In resource limited settings like Bangladesh, it is crucial to understand the factors that influence survival following an RTA in order to develop effective prevention strategies and improve patient outcomes. Therefore, this study aims to determine the 30 day survival rate and identify predictors of survival among adult RTA victims treated at a tertiary care hospital in Bangladesh. The observational study will be carried out at Emergency and casualty department of Dhaka Medical College Hospital (DMCH) between October 2025 and March 2026. A total of 204 adults (≥18 years) presenting to the hospital's Casualty Department with RTA related injuries will be included. Informed written consent will be obtained from each patient or their legal guardian prior to enrollment. Data will be collected through structured face to face interviews, review of hospital records, and follow up on the 30th day of accident. The follow-up will be conducted either in person or by telephone. Variables will include patient demographics, accident circumstances, admission characteristics, injury pattern and severity, pre-hospital care, clinical condition at admission, hospital management provided, and treatment outcome. All data will be analyzed using SPSS version 25.0. Kaplan-Meier analysis will estimate survival probabilities, while Cox proportional hazards regression will be used to identify independent predictors of mortality. The findings of this study are expected to generate context-specific, evidence-based insights for strengthening trauma care protocols, gap related to emergency handling of the RTA patients, enhancing pre-hospital emergency services, and informing policy decisions aimed at reducing preventable RTA-related mortality and morbidity in Bangladesh.

DETAILED DESCRIPTION:
Study Rationale:

Acne scars, notably atrophic scars, pose significant cosmetic and psychological concerns. Standard treatments include fractional lasers and microneedling-based interventions; however, rigorous comparative data in real-world clinical settings remain scarce. Recent evidence suggests ablative fractional CO2 laser and PRP-enhanced microneedling offer notable benefits. This split-face design allows direct comparison of efficacy, safety, and patient satisfaction between the modalities among Bangladeshi patients.

Study Design:

Type: Phase 3, open-label, randomized, split-face, comparative clinical trial

Planned Sample Size: 116 participants

Setting: Department of Dermatology, Dhaka Medical College Hospital, Bangladesh

Duration: April 2025 to March 2026

Randomization: Side of face assigned to either intervention via coin toss

Blinding: Open-label; outcome assessment by independent dermatologist blinded to intervention side

Eligibility Criteria:

Inclusion:

Age >18 years

Both sexes

Grade 2-4 acne scarring (Goodman & Baron qualitative grading)

Equal baseline scar grades on both facial halves

Atrophic scars only (no active acne)

Exclusion:

History of keloidal tendency

Bleeding or platelet disorders

Major surgery in past 6 months

Active facial infection (e.g., herpes, folliculitis)

HIV, hepatitis B surface antigen (HBsAg), or chronic illness

Pregnancy

Interventions:

Ablative Fractional CO2 Laser:

Pre-treatment: 2.5% lidocaine + 2.5% prilocaine cream (45 minutes), antiseptic cleansing

Device: SmartXide DOT Fractionated CO2 Laser (15 W, 800 μm spacing, 600 µs dwell, stack 2)

Three sessions, one month apart

PRP with Microneedling:

Pre-treatment: 2.5% lidocaine + 2.5% prilocaine cream (2 hours), antiseptic cleansing

PRP Preparation: 8 mL blood with double spin centrifugation to yield 2 mL PRP, platelet count verified

Intradermal PRP injection (nappage technique), followed by dermapen microneedling (1.5 mm depth, 12-needle cartridge, 4-directional passes)

Three sessions, one month apart

Follow-up and Data Collection:

Baseline, day 30, day 60, final (day 90 post first session)

Outcome measures collected via clinical assessments, standardized photographs, patient questionnaires, and independent dermatologist review

Adverse events monitored throughout

Outcome Measures:

Primary:

Change in Goodman & Baron quantitative and qualitative acne scar grades at 90 days

Secondary:

Independent dermatologist evaluation (10-point VAS, categorized for analysis)

Patient satisfaction (5-point Likert scale)

Frequency and type of adverse events/side effects

Subgroup analyses by scar severity, skin type, and sex

Statistical Analysis:

All analyses by intention-to-treat

Continuous data: Paired t-tests (within-group), independent t-test or Mann-Whitney U (between modalities)

Qualitative grades: McNemar's test (within-group), chi-square (between modalities)

Categorical responses (dermatologist VAS, satisfaction, side effects): chi-square or Fisher exact

95% confidence intervals, significance level 0.05

Safety Monitoring:

Data and Safety Monitoring Board (DSMB) of independent experts

GCP compliance and interim reviews

Adverse event reporting follows national and institutional guidelines

Ethical Considerations:

Written informed consent (Bengali/English)

Withdrawal permitted at any time without detriment to care

Confidential data handling in accordance with local regulations

Institutional ethics committee approval obtained

Keywords:

Acne scars, fractional CO2 laser, platelet-rich plasma, microneedling, randomized trial, Bangladesh, split-face, dermatology, Goodman and Baron, patient satisfaction, safety

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* Both male and female sex
* Patients with grade 2 to grade 4 acne scars, classiﬁed on the basis of Goodman's Qualitative classiﬁcation.
* Patient with equal Goodman's Qualitative scores on both halves of the face.
* No active acne lesions.
* Patients with atrophic scars only.

Exclusion Criteria:

* Positive history of keloidal tendency.
* Positive history of bleeding or platelet disorder.
* Positive history of major surgery in past 6 months.
* Presence of any acute infection on face like, herpes, folliculitis.
* Patients of HIV, HBsAg, or any chronic illness.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Goodman and Baron Acne Scar Grading (Quantitative and Qualitative) | Day 30 (prior to Session 2), Day 60 (prior to Session 3), and at the final follow-up visit on Day 150
  Improvement in acne scars will be assessed using the Goodman and Baron quantitative global acne scarring grading system and qualitative global acne scarring grading system.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhala Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) from this study. This decision is based on institutional policy, local regulatory considerations, and the need to protect participant confidentiality. De-identified data may be considered for sharing in the future upon appropriate request and with approval from the study's ethical review committee, but no prospective data sharing plan is in place at present.